CLINICAL TRIAL: NCT04486703
Title: Effect of Physical Therapy Rehabilitation Program Combined With Music on Pediatric With Lower Limb Burn: a Twelve-week Randomized Controlled Study
Brief Title: Physical Therapy Rehabilitation Program Combined With Music on Pediatric With Lower Limb Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6m8
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Lower Limb Burn
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with music group (Experimental): physical therapy program combined with music therapy
  Interventions: Other: Exercise with music
- Exercise group (Experimental): physical therapy program without music
  Interventions: Other: Exercise with music

INTERVENTIONS:
Other: Exercise with music — physical therapy program combined with music therapy 15 min, 3 times weekly for 12 weeks.

SUMMARY:
The purpose of the current study was to evaluate the effect of physical therapy rehabilitation program combined with music therapy on pediatric with lower limb burn. Methods. A twelve-week randomized controlled study including thirty lower limb pediatric burned patients who randomly divided into two groups, Group(A) received physical therapy rehabilitation program combined with music therapy in addition to routine medical care while Group (B) received physical therapy rehabilitation program without music therapy. Pain was assessed by visual analogue scale (VAS) and range of motion (ROM) was assessed by goniometer, and gait assessed by GAIT Rite. Assessment was carried before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Lower limb 2nd degree burn since 6 weeks
* Burn affect skin around ankle and knee joint,
* Both sex, age ranged between 10 to 15 years old
* Patients have sufficient cognition and education enough to understand the requirements of this study

Exclusion Criteria:

* All patients with age more than 15 years or less than 10 years
* Patients with hearing problems
* Acute viral diseases, acute tuberculosis, mental disorders
* Those with pace makers, diabetics, cardiac, renal patients
* Patients with genetic disease
* 3rd degree burn and 1st degree bum

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
pain in the lower limb | 12 weeks
  Visual analogue scale for pain assessment ,zero indicates no pain ten indicates maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided